CLINICAL TRIAL: NCT05097690
Title: Psychological Autopsy: An Investigation to Explore Antecedents, Sequelae and Causes of Case Control Suicide Equivocal Behavior
Brief Title: Case Control Psychological Autopsy of Suicide
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tamkeen Saleem (Other)
Collaborators: University of Leicester (Other); University of Warwick (Other); The American Association of Suicidology (Unknown)
Responsible Party: Sponsor-Investigator, Tamkeen Saleem, Assistant Professor, International Islamic University, Islamabad
Organization: International Islamic University, Islamabad (Other)
Other Study IDs: AAS-ATV-PAS
Record Dates: First submitted 2021-09-25; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Suicide; Fatal Suicide; Non Fatal Suicidal Behavior
Keywords: Cases; Controls
MeSH Terms: conditions — Suicide; Suicide, Completed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Case (Fatal Suicide)
- Control: Control (Non-Fatal Suicidal Behavior)

SUMMARY:
Suicide is a leading cause of death worldwide, and identifying risk factors has been considered as the key initiative of suicide prevention. Considering that, the study aimed to explore the factors leading towards suicide in Pakistan through Case-Control Psychological Autopsy of Suicide. Also, the study aimed to Translate, Adapt and Validate American Association of Suicidology (AAS) Semi-Structured Interview for Psychological Autopsy (Generic Version, 2018).

ELIGIBILITY:
Inclusion Criteria:

* The age of the deceased by suicide and living controls will range from 10 to 35 years.
* The key informants will be of 18 years of age and above without any learning
* disability.
* The key informants will be a close family member or immediate friend.
* Only suicides took place in 2019 to September 2021.

Exclusion Criteria:

* If contact was deemed to pose a risk to the safety of the researcher (likely intoxication; history of or potential for violence).
* Informants who are not willing to give written informed consent will be excluded from the study.
* Informants who are taking any psychological help in the past and present will be excluded from the study.

Ages: 10 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases are those individuals who died by suicide and the controls include individuals who survive after attempting suicide.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2022-02-25 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
The Semi-structured Interview for Psychological Autopsy | Upto 6 months
  American Association of Suicidology Semi-Structured Interview for Psychological Autopsy

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tamkeen Saleem, PhD, Study Chair — International Islamic University, Islamabad, Pakistan; Dr Michelle O'Reilly, PhD, Study Chair — University of Leicester and Leicestershire Partnership NHS Trust; Dr Domenico Giacco, PhD, Study Chair — Warwick Medical School, University of Warwick
Locations (1):
- International Islamic University, Islamabad Pakistan, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No